CLINICAL TRIAL: NCT06504758
Title: The Effects of Breathing Exercises and Postural Exercises Via Telerehabilitation on Respiratory Parameters, Posture, and Quality of Life in Young Adults With Asthma.
Brief Title: The Effects of Breathing Exercises and Postural Exercises in Young Adults With Asthma.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Elif Develi, Physiotherapist, Yeditepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IrmakC
Record Dates: First submitted 2024-07-04; First posted 2024-07-17 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Asthma
Keywords: Asthma; Young Adults; Breathing Exercises; Postural Exercises; Quality of Life; Posture; Asthma Control; Telerehabilitation; Oxygen Saturation; Respiratory Rate per Minute
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental): 12 young adults patients diagnosed with asthma.
  Interventions: Other: Breathing Retraining Program; Other: Postural Exerises Program (Stretching and Strengthening Exercises)

INTERVENTIONS:
Other: Breathing Retraining Program — * 1st to 5th week - Breathing Retraining 10 repetitions (Pursed Lip Breathing, Diaphragmatic Breathing)
  * Two days / a week The total duration of 5 weeks.
Other: Postural Exerises Program (Stretching and Strengthening Exercises) — * TheraBand® or Free Weight
  * 1st week - neck isometrics, chin tuck, SCM - upper trapezius - pectoral major stretching, scapular retraction without weight, rowing with yellow TheraBand®, wall squat / mini squat (5 repetitions - 15 second hold for stretching exercises, 10 repetitions for strengthening exercises)
  * 2nd and 3rd week - same exercises (5 repetitions - 15 second hold for stretching exercises, 15 repetitions for strengthening exercises)
  * 4th and 5th week - same exercises (10 repetitions - 15 second hold for stretching exercises, 20 repetitions for strengthening exercises)
  * Two days / a week,The total duration of 5 weeks

SUMMARY:
The aim of this study was to investigate the effects of breathing exercises and postural exercises via telerehabilitation on respiratory parameters, posture, and quality of life in young adults with asthma.

DETAILED DESCRIPTION:
12 young adult (18-25 years old) individuals diagnosed with asthma participated in our study (all female). All of the participants are University students.

Participants included in the study were evaluated with Asthma Control Test, Mini Asthma Quality of Life Questionnaire, International Physical Activity Questionnaire (short form) via Google Forms; Sit to Stand Test, Respiratory Rate per Minute and Oxygen Saturation were assessed at Yeditepe University Physiotherapy and Rehabilitation Laboratory both at baseline and at the end of the 5th week. Breathing and postural exercises were given to the participants for the duration of 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation in research.
* Patients in young adults (18-26 years old)
* Stable asthma.
* Modified Medical Counsel Research Dyspnea Test (mMRC) is 2 and above
* To stay consistent with an exercise program.

Exclusion Criteria:

* Being younger than 18 years old.
* Patients with severe asthma.
* Modified Medical Counsel Research Dyspnea Test (mMRC) is below 2

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-07-24 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
Mini - Asthma Quality of Life Questionnaire (AQLQ) | 5 weeks
  It is a test that measures health related quality of life in adults.
New York Posture Scale | 5 weeks
  There are 13 body alignment sections to general postural alignment. Includes posterior views of the head, shoulders, spine, hips, feet, and arches, and lateral (left side) views of the chest, shoulders, upper back, torso, abdomen, and lower back. Ratings were given as 5 (correct posture), 3 (minor deviation), or 1 (minor deviation).
Asthma Control Test | 5 weeks
  It is a questionnaire that consists of 5 topics referring to the daytime and nocturnal symptoms of past 4 weeks which are activity limitation, shortness of breath, awaking due to asthma symptoms, reliever medication and global judgment of asthma.
International Physical Activity Questionnaire - Short Form (IPAQ-SF) | 5 weeks
  It aims to evaluate physical activity across different nations in adults aged 18-65 years.
Oxygen Saturation | 5 weeks
  It is important to monitor current oxygen saturation due to the nature of oxygen consumption in the body.
Respiratory Rate Per Minute | 5 weeks
  The normal value of respiratory rate is roughly 12-16 breaths per minute.
Sit to Stand Test | 5 weeks
  Quadriceps muscle endurance will be evaluated with this test.

CONTACTS AND LOCATIONS:
Overall Officials: Irmak Sıla Çetinel, Principal Investigator — Yeditepe University; Elmas Teker, Principal Investigator — Yeditepe University; Beyda Ceyran, Principal Investigator — Yeditepe University
Locations (1):
- Yeditepe University, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No